CLINICAL TRIAL: NCT04493736
Title: CAMPUS Expanded "Classification and Assessment of Mental Health Performance Using Semantics Expanded"
Acronym: CAMPUS-E
Status: Recruiting | Type: Observational
Sponsor: Clarigent Health (Industry)
Responsible Party: Sponsor
Other Study IDs: Clarigent 104-2020
Record Dates: First submitted 2020-07-15; First posted 2020-07-30 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Suicide; Suicidal; Suicide, Attempted; Suicidal Ideation; Depression; Anxiety; Aggression; Trauma, Psychological
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicidal Ideation; Depression; Anxiety Disorders; Aggression; Psychological Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Audio recorded voice samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case: Any person receiving services from a mental health provider who is able to either consent or for whom parental consent is able to be obtained.
  Interventions: Behavioral: MHSAFE app recording

INTERVENTIONS:
Behavioral: MHSAFE app recording — Participants are asked a series of questions to elicit their feelings and emotions as part of an audio recorded interview along with their normal therapy session.

SUMMARY:
Open enrollment study to collect data for the optimization of machine learning models for use in an app for the early detection of mental health and suicidal risk.

ELIGIBILITY:
Inclusion Criteria:

* Currently a client receiving services from a MHP at a school or outpatient setting, or at a college/university counseling center
* Age ≥ 8 years old
* Able to provide informed consent, parental permission or assent
* English as a primary language

Exclusion Criteria:

* Participants with communication disorders (linguistic or articulation)
* Any minor participants for whom parental or legal guardian consent cannot be obtained.
* Any adult participant for whom Legal Authorized Representative (LAR) consent cannot be obtained.
* History of any other serious medical or psychiatric condition that would interfere with the ability of the patient to complete the study or would make it ethically unfeasible to enroll them
* Participants with an intellectual and / or neurocognitive disability that the MHP deems a barrier to participation
* Any participant, who at the discretion of the MHP, should not be enrolled

Ages: 8 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study employs a cohort design, using open and rolling recruitment of MHP participants at multiple locationssites nationally. We will recruit from mental health therapy practices, schools (using school based MHPs), community mental health agencies, or colleges/universities (counseling centers). Participating MHPs will begin enrolling client participants after completing the online protocol training and brief human subject's protection training. Recruitment will continue on a rolling basis until 2000 client participants have been enrolled and 6000 sessions have been recorded.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Detection of Mental Health State | 1 year
  Optimize machine learning models will detect the presence of a mental state as evidenced by scores on standardized tests and clinical assessment.

SECONDARY OUTCOMES:
Demonstrate the Usability of the platform | 1 year
  Demonstrate the usability of the MHSAFE recording platform and the dashboard output in different settings, including outpatient community mental health settings, schools (K-12), colleges/universities, and residential mental health facilities.

CONTACTS AND LOCATIONS:
Locations (1):
- Clarigent Health, Mason, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided